CLINICAL TRIAL: NCT01159561
Title: Phase 1 Study to Evaluate the Safety and Immunogenicity of the Western Equine Encephalitis (WEE) Vaccine, Inactivated, TSI-GSD 210, Lot 3-1-92, In Healthy Adults
Brief Title: Western Equine Encephalitis Vaccine, Inactivated
Acronym: WEE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A-15812; USAMRIID FY09-02 (Other: IRB)
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Virus
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccinated (Experimental): Western Equine Encephalitis Vaccine, Inactivated, TSI-GSD 210, Lot 3-1-92, administered in 0.5 mL doses subcutaneously in the upper outer aspect of the triceps in a 3-dose primary series (Days 0, 7, and 28) with a mandatory boost (Day 180)
  Interventions: Biological: Western Equine Encephalitis Vaccine

INTERVENTIONS:
Biological: Western Equine Encephalitis Vaccine — Subject will be vaccinated with 0.5 mL of reconstituted WEE vaccine, inactivated, TSI-GSD 210 (Lot 3-1-92) subcutaneously in the upper outer aspect of the deltoid region.

SUMMARY:
This study is designed to determine the safety and immunogenicity of WEE Vaccine Lot number 3-1-92.

DETAILED DESCRIPTION:
Study Objectives:

Primary: To assess safety of the Western Equine Encephalitis (WEE) Vaccine, Inactivated, TSI-GSD 210, lot 3-1-92.

Secondary: To evaluate immunogenicity of the Western Equine Encephalitis (WEE) Vaccine, Inactivated, TSI-GSD 210, lot 3-1-92.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years of age
* In good health as determined by pertinent medical history, brief physical exam, vital signs, and clinical safety laboratory evaluations
* Female: has a negative urine pregnancy test and is willing to use reliable form of contraception for the study duration
* Negative HIV antibody screen, seronegative for HBsAg and Hepatitis C antibody
* WEE, EEE, VEE, and CHIK PRNT80<1:10
* Ability to comprehend abnd a willingness to sign an informed consent, which includes the HIPAA and a separate HIV consent form
* Be willing to comply with all follow-up visits, testing, and AE reporting

Exclusion Criteria:

* Participant in the USAMRIID SIP
* Receipt of any other vaccine or investigational; drug within 30 days prior to study entry
* Anticipates receipt of other vaccines for the duration of the study (influenza vaccination will be permitted but not within 28 days of WEE vaccination
* Acute of chronic medical conditions, medications, or dietary supplements that, in the PI's opinion, would impair the subject's ability to respond to vaccination
* Hypersensitivity to any vaccine
* Allergic to any vaccine component: Human serum albumin, Neomycin
* Receipt of or anticipates receipt of blood products during the study
* Female: Pregnant or breastfeeding
* Clinically significant abnormal laboratory tests (generally greater than or equl to 2 times the upper limit of normal as determined by the PI)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Subjects Reporting Adverse Events by Vaccination and Sex | 28 days following each vaccination

SECONDARY OUTCOMES:
Immunogenicity | Baseline and multiple dates throughout study
  The primary endpoint used to measure immunogeniciyt of the WEE vaccine, the 80% plaque-reduction neautralization titer (PRNT 80), will be evaluated for subjects in the per protocol population.
  The secondary endpoint will be GMT, with 95% CI, of the PRNT 80 for WEE-specific antibodies at each scheduled timepoint.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B Reisler, MD, Principal Investigator — USAMRIID Medical Division
Locations (1):
- Clinical Research Unit, Division of Medicine, USAMRIID, Fort Deterick, Maryland, United States

REFERENCES:
- [Derived] Keshtkar-Jahromi M, Reisler RB, Haller JM, Clizbe DP, Rivard RG, Cardile AP, Pierson BC, Norris S, Saunders D, Pittman PR. The Western Equine Encephalitis Lyophilized, Inactivated Vaccine: An Update on Safety and Immunogenicity. Front Immunol. 2020 Nov 9;11:555464. doi: 10.3389/fimmu.2020.555464. eCollection 2020. PMID 33240257